CLINICAL TRIAL: NCT02038439
Title: Multifaceted Online Interventions to Increase the Quantity and Quality of Searching for Current Best Evidence to Answer Clinical Questions
Brief Title: Multifaceted Online Interventions to Increase Clinicians Searching of Current Best Evidence to Answer Clinical Questions
Acronym: MPFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: FRN86465
Record Dates: First submitted 2014-01-15; First posted 2014-01-16 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Physicians Evidence Retrieval Skills
Keywords: Evidence-Based Medicine; Evidence Retrieval; Knowledge Translation; Medical Education

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Interventions: A + B + C (Experimental): See Interventions Description. In this arm, clinicians will be offered all 3 online interventions combined:
  * Intervention A - Online Clinical Questions Recorder
  * Intervention B - Online Evidence Retrieval Coach
  * Intervention C - Online Audit and Feedback
  Interventions: Behavioral: Intervention A - Online Clinical Questions Recorder; Behavioral: Intervention B - Online Evidence Retrieval Coach; Behavioral: Intervention C - Online Audit and Feedback
- Interventions A + B (Experimental): See Interventions Description. In this arm, clinicians will be offered the 2 following interventions combined:
  * Intervention A - Online Clinical Questions Recorder
  * Intervention B - Online Evidence Retrieval Coach
  Interventions: Behavioral: Intervention A - Online Clinical Questions Recorder; Behavioral: Intervention B - Online Evidence Retrieval Coach
- Interventions A + C (Experimental): See Interventions Description. In this arm, clinicians will be offered the 2 following online interventions combined:
  * Intervention A - Online Clinical Questions Recorder
  * Intervention C - Online Audit and Feedback
  Interventions: Behavioral: Intervention A - Online Clinical Questions Recorder; Behavioral: Intervention C - Online Audit and Feedback
- Interventions B + C (Experimental): See Interventions Description. In this arm, clinicians will be offered the 2 following online interventions combined:
  * Intervention B - Online Evidence Retrieval Coach
  * Intervention C - Online Audit and Feedback
  Interventions: Behavioral: Intervention B - Online Evidence Retrieval Coach; Behavioral: Intervention C - Online Audit and Feedback
- Intervention A alone (Experimental): See Interventions Description. In this arm, clinicians will be offered only the following intervention:
  * Intervention A - Online Clinical Questions Recorder
  Interventions: Behavioral: Intervention A - Online Clinical Questions Recorder
- Intervention B alone (Experimental): See Interventions Description. In this arm, clinicians will be offered only the following intervention:
  * Intervention B - Online Evidence Retrieval Coach
  Interventions: Behavioral: Intervention B - Online Evidence Retrieval Coach
- Intervention C alone (Experimental): See Interventions Description. In this arm, clinicians will be offered only the following intervention:
  * Intervention C - Online Audit and Feedback
  Interventions: Behavioral: Intervention C - Online Audit and Feedback
- No intervention (No Intervention): In this arm, clinicians will be offered non of the 3 online interventions, but will just be using the usual features of the search engine available to all users.

INTERVENTIONS:
Behavioral: Intervention A - Online Clinical Questions Recorder — Clinicians allocated to this intervention will receive access to an online recorder for the clinical questions at the point of care. The recorder is accessible across a wide range of devices including phones, tablets, and desktop computers.
  Arms: Intervention A alone; Interventions A + B; Interventions A + C; Interventions: A + B + C
Behavioral: Intervention B - Online Evidence Retrieval Coach — Clinicians allocated to this intervention will receive online guidance, embedded in the MPFS search engine, in the form of short videos, animations, demos and tips and tricks regarding evidence retrieval.
  Arms: Intervention B alone; Interventions A + B; Interventions B + C; Interventions: A + B + C
Behavioral: Intervention C - Online Audit and Feedback — Clinicians allocated to this intervention will receive feedback on their current search performance compared to their peers, both online when using MPFS as well as by e-mail.
  Arms: Intervention C alone; Interventions A + C; Interventions B + C; Interventions: A + B + C

SUMMARY:
Translation of new knowledge from research into evidence-informed health care is a shared obligation of the clinical and the scientific communities. Unfortunately, studies of quality of care continue to show that this goal is substantially unrealized. One main barrier is lack of quick and easy identification, appraisal and synthesis of current best evidence. Clinicians' information have 5 to 8 questions about individual patients per daily shift, but face a large volume of 3000 articles published every day, accessible in many scattered resources.

To address theses problems, McMaster's Health Information Research Unit (Hamilton, Ontario, Canada) has developed and implemented "McMaster Premium LiteratUre Service Federated Search" (MPFS), an online search engine that provides a unique 1-stop search and organized access to current best evidence in daily practice. However additional barriers need to be overcome for clinicians to actually search and use this evidence in their practice. Theses include logistical barriers (time constraints, forgotten questions), as well as educational barriers (eg, lack of awareness of the "architecture" of evidence, limited searching skills, and lack of reference standards among peers for finding best evidence).

This randomized trial seeks to test 3 innovative online interventions among clinicians registered to MPFS to overcome these barriers and increase the quantity and quality of searching for current best evidence to answer clinical questions. These interventions build on effective models for the teaching of clinical skills at the point of care, so that clinicians are facilitated in using the search engine as a clinical tool, and perceive evidence retrieval skills as true clinical skills.

DETAILED DESCRIPTION:
1. Rationale & Objectives

   One main barrier to achieving evidence-informed care by clinicians is lack of quick and easy identification, appraisal and synthesis of current best evidence. Clinicians' information needs are considerable - but about 3000 articles are published in Medline every day. Numerous evidence-based resources have been developed to filter and process the evidence, but although increasingly used by clinicians, each offer a fragmented and scattered view of information, and none provides comprehensive topic coverage or satisfactory updating.

   To address theses problems, McMaster's Health Information Research Unit (Hamilton, Ontario, Canada) has developed and implemented "McMaster Premium LiteratUre Service Federated Search (MPFS)", an online search engine that provides a unique 1-stop search and organized access to current best evidence in daily practice. MPFS provides both alerts to users about new research in their chosen disciplines, and a novel federated search function, with the particular feature of organizing information according to the "pyramid of evidence-based resources", with the most clinically applicable evidence at the top. Thus MPFS simultaneously retrieves evidence from Studies ("Medline", both filtered and unfiltered, at the bottom), then Systematic reviews; Synopses of studies and systematic reviews (selected for methodological rigor and clinical relevance), and, at the top level, online widely used Summaries (e.g."Best Practice").

   Combining features of the current best evidence-based resources is not enough to increase access and use of current best evidence, as shown by the relatively low utilization of searching features among the hundreds of clinicians currently registered at McMaster University and using the alerting system. Additional well-known barriers that need to be overcome include logistical barriers (time constraints, forgotten questions, and simplicity of using one single albeit limited resource), as well as educational barriers (eg, lack of awareness of the "architecture" of evidence and limits of other single resources, lack of knowledge and experience of what federated searches can offer, limited searching skills, and lack of reference standards among peers for finding best evidence).
2. Hypothesis

   This trial seeks to test 3 innovative online interventions among clinicians registered to MPFS to overcome these barriers and increase the quantity and quality of searching for current best evidence to answer clinical questions. These interventions build on effective models for the teaching of clinical skills at the point of care, so that clinicians are facilitated in using the search engine as a clinical tool, and perceive evidence retrieval skills as true clinical skills.
3. Methods

   1. Study design: Randomized Factorial Controlled Trial.
   2. Setting and Participants: The trial will be conducted among postgraduate and faculty MD registered in MPFS and working in the teaching hospitals and clinics of McMaster University (see eligibility criteria below)
   3. Participating clinicians will be randomized to 3 online interventions (see description below) in a factorial design (A x B x C), whose permutation results in 8 allocation arms (A+B+C, A+B, A+C, B+C, A, B, C, no intervention, see details below)
   4. Randomization: will be computer-generated, stratified training level (post-graduate MD, faculty MD), and baseline frequency of searching for evidence on MPFS. Registrants will be randomly allocated to each study arms. Allocation will be concealed from research staff.
   5. Blinding and control group: Although participants cannot be blinded to the interventions, they will not be told of the different features offered, and all will receive usual searching features of MPFS.
   6. Primary and secondary outcomes (see below).

ELIGIBILITY:
Inclusion Criteria:

* All postgraduate and faculty physicians currently registered for more than one month in the MPFS search engine,
* and working in the teaching hospitals and clinics of the Faculty of Health Sciences, McMaster University, Hamilton, Ontario.

Exclusion Criteria:

* Registrants that are no longer working or training at McMaster University,
* Registrants that never logged in MPFS during the last 12 months counting back from the beginning of the trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 908 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Utilization of evidence-based resources on MPFS as measured by rate of searches/month/user | 6 months
  Each clinician participating in the trial has a personal online account in MPFS. When they are signed on their account, the system continuously tracks their searches and utilization of individual resources. We will record their utilization over the full duration of the trial (6 months) and analyze it in the end.

SECONDARY OUTCOMES:
Utility (satisfaction in meeting users' information needs) as assessed by the Impact Assessment Measure questionnaire | 6 months
  This Impact Assessment Measure questionnaire will be sent to clinicians after a random sample of searches and completed online for a random sample of searches.
Use (application of evidence in practice) as assessed by the Impact Assessment Measure questionnaire | 6 months
  This Impact Assessment Measure questionnaire will be sent to clinicians after a random sample of searches and completed online for a random sample of searches.
Perceived Usefulness in patient care and outcomes as assessed by the Impact Assessment Measure questionnaire | 6 months
  This Impact Assessment Measure questionnaire will be sent to clinicians after a random sample of searches and completed online for a random sample of searches.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Agoritsas, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Seguin A, Haynes RB, Carballo S, Iorio A, Perrier A, Agoritsas T. Translating Clinical Questions by Physicians Into Searchable Queries: Analytical Survey Study. JMIR Med Educ. 2020 Apr 20;6(1):e16777. doi: 10.2196/16777. PMID 32310137
- [Derived] Agoritsas T, Iserman E, Hobson N, Cohen N, Cohen A, Roshanov PS, Perez M, Cotoi C, Parrish R, Pullenayegum E, Wilczynski NL, Iorio A, Haynes RB. Increasing the quantity and quality of searching for current best evidence to answer clinical questions: protocol and intervention design of the MacPLUS FS Factorial Randomized Controlled Trials. Implement Sci. 2014 Sep 20;9:125. doi: 10.1186/s13012-014-0125-9. PMID 25239537
- See also: online MPFS search engine — http://plus.mcmaster.ca/MacPLUSFS/